CLINICAL TRIAL: NCT01533909
Title: Development of a Screening Tool to Detect and Stage Cachectic Cancer Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54035
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2012-03

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The blood sample that will be collected is part of the routine hospital assessment. The biomarkers that will be measured are albumine, creatine, CRP, hemoglobin and Lactate dehydrogenase (LDH).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients: As this is not an intervention study there is only one cohort. Patients that will be included and excluded are described in the eligibility section.

SUMMARY:
The aim of the study is to develop a screenings tool that will enable hospital nurses to detect and stage cancer cachectic patients. The early detection and staging of cancer cachexia will assist the oncology team in providing the cachectic cancer patient tailor-made patient care.

DETAILED DESCRIPTION:
In this cross-sectional study, the participants will complete 4 times a set of questionnaires and measurements. The data that will be collected is:

age; sex; height; weight; type of tumour; classification of malignant tumours (TNM); progression of tumour and used therapy; blood sample to analyse albumin, creatine, hemoglobin, LDH and CRP; use of parental nutrition; dietary assessment; use of nutritional supplements; Quality of Life by using the EORTC-QlQ; Subjective Global Assessment; presence of Percutaneous endoscopic gastrostomy; use of enteral or parenteral nutrition; body composition based on a Bio Impedance Assessment; hand grip strength and mid upper arm circumference. Based on all these data points a easy to use tool/score for a hospital setting will be created. During the first assessment the measurements will be done in the morning and the evening to test the reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* New Diagnosed Patients With Primary Head and Neck Cancer Neoplasms
* New Diagnosed Patients With Metastatic Pancreatic Neoplasms
* New Diagnosed Patients With Metastatic Colonic Neoplasms

Exclusion Criteria:

* Patients With Other Primary Neoplasms
* Patients Already in Therapy
* Patients With Non-metastatic Colonic or Pancreatic Neoplasms

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from which the groups or cohorts will be selected (e.g., primary care clinic, community sample, residents of a certain town). (Limit: 1000 characters)
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Nutritional Assessment | 4 times in 6 months
  Patient-Generated Subjective Global Assessment Instrument is a measure for the nutritional status of the participants. The final score of this instruments devides participants into three categories: well-nourished, moderately nourished or suspected malnourished.

SECONDARY OUTCOMES:
Quality of Life | 4 times in 6 months
  The EORTC-QlQ questionnaire will be used to assess the quality of life of the participants.
Anthropometric measurements | 4 times in 6 months
  Mid-upper arm circumference will be measured to have an idea of the muscle mass.
  Hand Grip Strength will be measured to obtain an idea of the muscle strength. Weight will be measured during every occasion. Question will be asked about weight loss during the last 6 months. Body composition will be measured by Bio-impedance assessment to obtain an indication of the fat-free mass.
  Changes of all these measurements will be monitored.
Markers of inflammation/metabolic disturbance | 4 times in 6 months
  Biomarkers will be selected as part of the routine hospital assessment. These markers are C-reactief proteïne, albumin, creatinin, hemoglobin and Lactate dehydrogenase (LDH). These markers are a measure of the nutritional status and are seen as markers for the catabolic state of cachectic cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Vergote, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Vlaams Brabant, Belgium